CLINICAL TRIAL: NCT03790566
Title: Comparison of Erector Spinae Plane Block With Transversus Abdominus Plane Block for Peri-operative Pain Management in Pediatric Open Pyeloplasty Cases
Brief Title: Erector Spinae Plane Block for Peri-operative Pain Management in Pediatric Open Pyeloplasty Cases
Acronym: ESPPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Collaborators: Aybike Onur Gonen (Unknown); Ayse Cigdem Tutuncu (Other); Kaya, Guner, M.D. (Individual); Rahsan Ozcan (Unknown)
Responsible Party: Principal Investigator, pinar kendigelen, Assoc. Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 72109855-604.01.01-53213
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia and Analgesia; Pediatrics; Urologic Surgical Procedures
Keywords: ESP block; TAP block; pyeloplasty; erector spina plane block; transversus abdominus plane block; flank incision; post-op analgesia; peri-op analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental): With the patient in lateral decubitus position (surgical side up), the transverse processes of T10-T12 vertebrae and erector spinae (ES) fascia are visualized 1-2 cm lateral to the vertebral spine using a linear ultrasound probe. A 22G peripheral block needle is introduced with in-plane technique under the ES muscle and local anesthetic solution (0.5 ml/kg 0.25% bupivacaine) is injected in this plane after a test injection with 0.5 ml of 0.9% NaCl solution to visualize opening of ESP.
  Interventions: Drug: Bupivacaine
- Transversus abdominus plane block (Active Comparator): With the patient in supine position, three layers of abdominal muscle are visualized using the linear ultrasound probe held with the long axis on the mid-axillary line above the iliac crest. 22G peripheral block needle is introduced in-plane into the fascia between the internal oblique and transversus abdominus muscles and local anesthetic solution (0.5 ml/kg 0.25% bupivacaine) is injected in this plane after a test injection with 0.5 ml of 0.9% NaCl solution to visualize opening of ESP.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.5 ml/kg 0.25% bupivacaine

SUMMARY:
Regional anesthesia decreases the need for intravenous analgesia in the peri-operative period. Erector spinae plane (ESP) and transversus abdominus plane (TAP) blocks are two common regional anesthesia techniques shown to be effective in open abdominal surgeries. We aim to compare effectiveness of ESP block with TAP block for peri-operative analgesia in pediatric open pyeloplasty patients with a flank incision.

DETAILED DESCRIPTION:
Regional anesthesia for effective post-operative pain management is a part of the pediatric Enhanced Recovery After Surgery (ERAS) protocol. Epidural anesthesia is the gold standard for analgesia for open abdominal surgeries, however difficulties in application and possible complications deter clinicians from utilizing this method. Safe and effective alternatives to epidural anesthesia has been a critical and popular focus of clinical research in recent years. Transversus abdominus plane (TAP) block is an alternative technique shown to be effective in pediatric open abdominal surgeries.

Erector spinae plane (ESP) block was described as an effective block for multi-dermatome pain after thoracic surgery. It is emerging as a safe and easy-to-perform alternative to epidural anesthesia for pelvic, abdominal and thoracic surgery.

During an open pyeloplasty, the flank incision goes through the transversus abdominus plane, where the local anesthetic is injected for TAP block. This may weaken the analgesic effect of the block. In the ESP block, local anesthetic diffuses cranio-caudally through the fascia of erector spinae muscles and the flank incision does not disturb this plane. We aim to compare the effectiveness of ESP block with TAP block in open pyeloplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class I, II or III
* Patients scheduled for elective open pyeloplasty surgery

Exclusion Criteria:

* Local anesthetic allergy or other contraindication to local anesthetic use
* Coagulation disorders
* History of chronic pain
* Patient/Family refusal
* History of scoliosis, spinae bifida, abdominal wall defect
* Past surgical procedures with abdominal wall incision
* Plan to extend the flank incision for additional surgical intervention

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-09-02 (Estimated); Study Completion 2019-09-25 (Estimated)

PRIMARY OUTCOMES:
Remifentanil need | During the operation
  Intraoperative remifentanil requirement as rescue analgesia
Post-operative analgesia need | 24 hours post-operatively
  Pain score is assessed with FLACC (Face, Legs, Activity, Cry, Consolability) scale. A score of 2, 3, 4 or 5 warrants for intravenous paracetamol need and a score of 6 and above warrants for intravenous tramadol

SECONDARY OUTCOMES:
Parental satisfaction with analgesia | 24 hours post-operatively
  Parents will be asked how satisfied they are with the patient's pain control: 1. Dissatisfied, 2. Partially satisfied 3. Satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Kendigelen, Assoc. Prof., Principal Investigator — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided